CLINICAL TRIAL: NCT04568512
Title: DNA Methylation Biomarker in Biliary Brush Sample for Diagnosis of Cholangiocarcinoma in Patients With Bile Duct Stricture
Brief Title: DNA Methylation Biomarker for Diagnosis of Cholangiocarcinoma in Patients With Bile Duct Stricture
Acronym: DNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 149/2559
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Cholangiocarcinoma; Biliary Stricture; DNA Methylation; Brush Cytology
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Brushed biliary samples from a known case of benign biliary stricture were sent for DNA Methylation Biomarker test and cell cytology
  Interventions: Diagnostic Test: Control
- Cholangiocarcinoma (Active Comparator): Brushed biliary samples from a known case of cholangiocarcinoma were sent for DNA Methylation Biomarker test and cell cytology
  Interventions: Diagnostic Test: Cholangiocarcinoma

INTERVENTIONS:
Diagnostic Test: Control — Brushed biliary samples from a known case of benign biliary stricture were sent for DNA Methylation Biomarker test and cell cytology
  Arms: Control
Diagnostic Test: Cholangiocarcinoma — Brushed biliary samples from a known case of cholangiocarcinoma were sent for DNA Methylation Biomarker test and cell cytology
  Arms: Cholangiocarcinoma

SUMMARY:
DNA methylation biomarker for diagnosis of cholangiocarcinoma in patients with bile duct stricture has high sensitivity and specificity compared with cytology from the brush specimens

DETAILED DESCRIPTION:
The methylation of HOXA1, NEUROG1 were used to determine cholangiocarcinoma from brushed biliary samples. However, the sensitivity and specificity of this test for cholangiocarcinoma is still required.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 year old
* Patients had biliary stricture from cholangiocarcinoma and benign stricture

Exclusion Criteria:

* Pregnancy
* Patient had other malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The methylation of HOXA1, NEUROG1 were determined in brushed biliary samples from patients with CCAs compared to those of nonmalignant bile duct stricture | 2 weeks
  Methylation index of biliary brush samples were analyzed.

SECONDARY OUTCOMES:
Sensitivity, specificity of DNA methylation for diagnosis of cholangiocarcinoma | 2 weeks
  Diagnostic accuracy of methylation index for diagnosis of cholangiocarcinoma was analyzed.
To compared sensitivity, specificity of DNA methylation with routine cytology of biliary brushed samples | 2 weeks
  Diagnostic accuracy of methylation index was compared to routine brush cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Varayu Prachayakul, Principal Investigator — Mahidol University
Locations (1):
- Faculty of medicine, Siriraj hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prachayakul V, Rugivarodom M, Nopjaroonsri P, Cheirsilpa K, Chang A, Kamolhan T, Boonyaarunnate T, Thuwajit C, Thuwajit P. Diagnostic power of DNA methylation markers suggestive of cholangiocarcinoma in ERCP-based brush cytology. Gastrointest Endosc. 2022 Jan;95(1):123-130.e1. doi: 10.1016/j.gie.2021.07.005. Epub 2021 Jul 12. PMID 34265285